CLINICAL TRIAL: NCT02439879
Title: Treatment With Alpha-lipoic Acid Over 16 Weeks in Type 2 Diabetic Patients With Symptomatic Polyneuropathy Who Responded to Initial 4-week High-dose Loading
Brief Title: Alpha Lipoic Acid for Treatment of Diabetic Neuropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Popular Autónoma del Estado de Puebla (Other)
Responsible Party: Principal Investigator, Hector Garcia-Alcala, Endocrinology professor, Universidad Popular Autónoma del Estado de Puebla
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPAEP25082009
Record Dates: First submitted 2015-05-04; First posted 2015-05-12 (Estimated); Results first posted 2016-03-02 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Thioctic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- alpha lipoic acid treatment (Active Comparator): After a decrease in the total symptoms score >3 points with 600 mg orally tid of alpha lipoic acid for 4 weeks patients were randomized to recieve for 16 weeks 600 mg orally once a day of alpha lipoic acid
  Interventions: Drug: Alpha lipoic acid
- alpha lipoic acid withdrawal (No Intervention): After a decrease in the total symptoms Score >3 points with 600 mg orally tid of alpha lipoic acid for 4 weeks patients were randomized to recieve for 16 weeks no treatment

INTERVENTIONS:
Drug: Alpha lipoic acid — Alpha lipoic acid 1800 mg PO divided in 3 doses for 4 weeks . If total symptoms score decreased >3 points patients received alpha lipoic acid 600 mg PO each day or no treatment for 16 weeks.
  Other Names: Thioctic acid; Thioctacid HR
  Arms: alpha lipoic acid treatment

SUMMARY:
Patients with diabetic neuropathy and total symptoms score(TSS) >7 points were invited to this open multicenter study. Patients were free of pain medications and severe diabetic complications .Patients started alpha lipoic acid (ALA)1800 mg for 4 weeks. Patients with a decrease >3 points in the TSS were randomly allocated to 600 mg of ALA (ALA group) or no medications (ALA withdrawal) for 16 weeks. In each visit investigators evaluated any change in the TSS and the necessity of rescue medication to control symptoms (mainly pain). At the end of the study investigators compared between ALA and ALA withdrawal groups TSS levels and the frequency of use of rescue medications. Physicians were free to manage glucose to maintain Hba1c close to the ADA target (HbA1c <7%).

DETAILED DESCRIPTION:
This trial was conducted in accordance with the Declaration of Helsinki and was approved by the ethics committee of Universidad Popular Autónoma del Estado de Puebla, Mexico. All participants provided a written informed consent. Type 2 diabetic patients (according to American Diabetes Association (ADA) criteria) with symptomatic diabetic sensorimotor polyneuropathy (DSPN) defined as the presence of neuropathic symptoms (pain, paresthesias, or numbness) were invited to participate in this open-label multicenter trial. Inclusion criteria were: total symptom score (TSS) >7 points, HbA1c<10%, and serum creatinine <2 mg/dl. Exclusion criteria were evidence of active cardiovascular disease, malignancy, or any other conditions causing neuropathic pain, use of analgesic, antidepressant, or antiepileptic drugs, or any other medication aimed to relief neuropathic pain. In addition, child-bearing female patients not using any effective birth control method and under surveillance of a board-certified gynecologist were excluded.

Phase 1. All patients meeting inclusion criteria received 600 mg of alpha lipoic acid (ALA) (Meda Pharma, Germany) orally tid, 30 min after each main meal for 4 weeks. During phase 1, no medication for relief of neuropathic pain was allowed. Each participating site was in charge to maintain glycemic control based on the investigator's judgment attempting that all patients were treated according to the american diabetes association (ADA) guidelines. All patients were seen once a week, and at each site visit, TSS was assessed along with a pill count to ensure drug adherence, presence of adverse events and, if needed, treatment adjustments to maintain glucose levels within the ADA targets. Patients with a TSS reduction >3 points by the end of phase 1 were selected to proceed with phase 2 of the study. Patients with a decrease <3 points in TSS or that used other neuropathic pain drugs were excluded from study phase 2.

Phase 2. Patients with a decrease of ≥3 TSS points after phase 1 were randomized to receive 600 mg of ALA orally qd for 16 weeks or ALA withdrawal. Patients were scheduled to visit the clinic every 2-3 weeks for TSS, monofilament and assessment. If needed, the patient was prescribed analgesic rescue medication which was monitored at each visit. Primary endpoint was the change in TSS in the two groups studied in phase 2 and the frequency of use of rescue medications Neurological examination was performed at baseline and after phase 1 and 2 including the monofilament test, vibration perception threshold (VPT), and ankle reflexes. A 10g nylon monofilament (Thio-Feel ® Meda Pharma, Germany) was applied to four anatomical sites in each foot (1st, 3rd and 5th metatarsal heads and plantar surface of distal hallux) as previously described (correct answer = 1 point, with a maximum of 4 points in each foot). Eight correct answers were considered normal, 1-7 correct answers indicated reduced monofilament sensation, while absent sensation was assumed if no answer was correct. VPT was evaluated using a 128-Hz tuning fork (Thio-Vib ®, Meda Pharma,Germany) applied bilaterally at the tip of the great toe. Responses were categorized as abnormal (no perception of vibration), present (examiner perceives vibration <10 seconds after patient reported disappearance of vibration perception) and reduced (examiner perceives vibration >10 sec after patient reported disappearance of vibration perception). Ankle reflexes were graded as normal, decreased, and absent

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients (according to American Diabetes Association (ADA) criteria)
* Symptomatic diabetic polyneuropathy
* Total Symptom Score (TSS) >7 points,
* HbA1c<10%,
* Serum creatinine <2 mg/dl.

Exclusion Criteria:

* Active cardiovascular disease
* Malignancy
* Any other conditions causing neuropathic pain
* Use of analgesic, antidepressant, or antiepileptic drugs, or any other medication aimed to relief neuropathic pain.
* Child-bearing female patients not using any effective birth control method and under surveillance of a board-certified gynecologist

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hector Garcia-Alcala, MD, Principal Investigator — Universidad Popular Autonoma del Estado de Puebla

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Papanas N, Ziegler D. Efficacy of alpha-lipoic acid in diabetic neuropathy. Expert Opin Pharmacother. 2014 Dec;15(18):2721-31. doi: 10.1517/14656566.2014.972935. Epub 2014 Nov 10. PMID 25381809
- [Result] Ziegler D, Papanas N, Vinik AI, Shaw JE. Epidemiology of polyneuropathy in diabetes and prediabetes. Handb Clin Neurol. 2014;126:3-22. doi: 10.1016/B978-0-444-53480-4.00001-1. PMID 25410210
- [Result] Brownrigg JR, de Lusignan S, McGovern A, Hughes C, Thompson MM, Ray KK, Hinchliffe RJ. Peripheral neuropathy and the risk of cardiovascular events in type 2 diabetes mellitus. Heart. 2014 Dec;100(23):1837-43. doi: 10.1136/heartjnl-2014-305657. Epub 2014 Aug 5. PMID 25095826
- [Result] Finnerup NB, Attal N, Haroutounian S, McNicol E, Baron R, Dworkin RH, Gilron I, Haanpaa M, Hansson P, Jensen TS, Kamerman PR, Lund K, Moore A, Raja SN, Rice AS, Rowbotham M, Sena E, Siddall P, Smith BH, Wallace M. Pharmacotherapy for neuropathic pain in adults: a systematic review and meta-analysis. Lancet Neurol. 2015 Feb;14(2):162-73. doi: 10.1016/S1474-4422(14)70251-0. Epub 2015 Jan 7. PMID 25575710
- [Result] Ziegler D, Buchholz S, Sohr C, Nourooz-Zadeh J, Roden M. Oxidative stress predicts progression of peripheral and cardiac autonomic nerve dysfunction over 6 years in diabetic patients. Acta Diabetol. 2015 Feb;52(1):65-72. doi: 10.1007/s00592-014-0601-3. Epub 2014 Jun 5. PMID 24898524
- [Result] Ziegler D, Low PA, Litchy WJ, Boulton AJ, Vinik AI, Freeman R, Samigullin R, Tritschler H, Munzel U, Maus J, Schutte K, Dyck PJ. Efficacy and safety of antioxidant treatment with alpha-lipoic acid over 4 years in diabetic polyneuropathy: the NATHAN 1 trial. Diabetes Care. 2011 Sep;34(9):2054-60. doi: 10.2337/dc11-0503. Epub 2011 Jul 20. PMID 21775755
- [Derived] Garcia-Alcala H, Santos Vichido CI, Islas Macedo S, Genestier-Tamborero CN, Minutti-Palacios M, Hirales Tamez O, Garcia C, Ziegler D. Treatment with alpha-Lipoic Acid over 16 Weeks in Type 2 Diabetic Patients with Symptomatic Polyneuropathy Who Responded to Initial 4-Week High-Dose Loading. J Diabetes Res. 2015;2015:189857. doi: 10.1155/2015/189857. Epub 2015 Aug 4. PMID 26345602

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Type 2 diabetic patients with symptomatic neuropathic symptoms from 3 medical clinics in Puebla city, Mexico (one private, 2 public) were invited direct by investigator to participate if they fulfill inclusion criteria and no exclusion criteria. First patient was included on January 8th 2010 and the last visit of one patient was on December 2010
Pre-assignment Details: All patients meeting inclusion criteria received 600 mg of alfa-lipoic acid orally tid for 4 weeks. Patients with a TSS reduction >3 points by the end of phase 1 were selected to proceed with phase 2 of the study. Patients with a decrease <3 points in TSS or who used other neuropathic pain drugs were excluded from study phase 2.
Period: Overall Study
Arm/Group | Alpha Lipoic Acid Treatment | Alpha Lipoic Acid Withdrawal
Started | 16 | 17
Completed | 16 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alpha Lipoic Acid Treatment | Alpha Lipoic Acid Withdrawal | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (10) | 59 (11) | 58.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 5 | 6 | 11
TSS [Mean (Standard Deviation); unit: units on a scale] — Total Symptoms Score TSS, which is a summation of the presence, severity,and duration of lancinating pain, burning pain, prickling, and asleep numbness. Each of these is a positive neuropathic sensory symptom. Scoring: total score 0-14.64. Any increase in the score means a worsening of symptoms
  units on a scale | 3.7 (1.97) | 3.23 (2.07) | 3.45 (2)

OUTCOME MEASURES:

1. Primary Outcome: Total Symptoms Score
Description: Total symptoms score is a summation of presence, severity, and duration of the four main positive neuropathic sensory symptoms: lancinating/stabbing pain, burning pain, paresthesia, and asleep numbness
Time Frame: 20 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Alpha Lipoic Acid Treatment | Alpha Lipoic Acid Withdrawal
Number analyzed (Participants) | 16 | 17
units on a scale | 2.5 (0.6) | 3.1 (0.8)
Statistical Analysis 1: Comparison: Alpha Lipoic Acid Treatment vs Alpha Lipoic Acid Withdrawal; All data were analyzed using the SPSS v16 statistical package software. To compare categorical variables, the chi2 test was used, and, for continuous variables,the T-test for independent or paired samples was applied.Data are expressed as percent values with 95% confidence intervals (CI) or mean ± SD or mean ± SEM; Test type: Superiority or Other; p < 0.05, paired t test

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Alpha Lipoic Acid Treatment | Alpha Lipoic Acid Withdrawal
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No